CLINICAL TRIAL: NCT00001103
Title: Cerebrospinal Fluid Human Immunodeficiency Virus-1 (HIV-1) and Cognitive Function in Individuals Receiving Potent Antiretroviral Therapy
Brief Title: HIV Levels in Cerebrospinal Fluid and Brain Function in Patients Receiving Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Neurologic AIDS Research Consortium (NARC) (Other)
Other Study IDs: ACTG 736; AACTG 736
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2006-05

CONDITIONS: Cognitive Disorders; HIV Infections
Keywords: Neuropsychological Tests; HIV-1; RNA, Viral; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — Cognitive Dysfunction; HIV Infections

SUMMARY:
The purpose of this study is to see whether anti-HIV drugs that reduce HIV in the blood also reduce HIV in the cerebrospinal fluid (CSF). CSF is the fluid found around the brain and spinal cord. This study also looks at whether reducing HIV in the CSF can help protect brain function.

HIV can be detected in the brain and CSF early in HIV disease. Anti-HIV drugs probably reduce HIV in the CSF. This may be important because other studies have suggested high CSF HIV levels may lead to some loss of brain function.

DETAILED DESCRIPTION:
HIV-1 RNA emerges in CSF early in the course of HIV disease. Studies have shown that high levels of HIV-1 RNA in CSF correlate with increased severity of dementia and worsened performance on neuropsychological tests. While combination antiretroviral treatments are potent suppressors of HIV-1 replication in plasma, the extent to which these treatments suppress viral replication in CSF is unknown. A few studies suggest that antiretroviral treatments can reduce HIV-1 RNA in CSF. However, since CSF is isolated from peripheral immune responses to HIV and antiretroviral treatment may not readily penetrate the compartment, researchers hypothesize the remaining virus will overcome the antiretroviral treatment to achieve high levels of viral replication again. This virologic failure is likely accompanied by decreased cognitive function. It is therefore critical to determine the ability of antiretroviral treatments to control HIV-1 replication in the CSF and the durability of that viral suppression.

Patients enrolling in one of several AACTG-sponsored potent antiretroviral therapy trials (a "parent" trial) may enter this study. [AS PER AMENDMENT 06/06/00: Patients already enrolled in an AACTG-sponsored study who are changing treatment due to virologic failure may also enter this study.] [AS PER AMENDMENT 11/15/01: Patients starting a new potent antiretroviral regimen as part of their clinical care, enrolling in a potent antiretroviral treatment trial, or changing potent antiretroviral therapy in clinical care or in an ongoing antiretroviral treatment trial because of virologic failure may enter this study.] Patients receive no treatment but undergo various procedures aimed at characterizing the effects of antiretroviral therapies on CSF viral load and cognitive function. Procedures include: 1) venipuncture to measure plasma HIV-1 RNA and DNA levels, CD4+ T cell count, and cytokine and immune activation markers associated with HIV-1 neurological disorders; 2) neuropsychological examinations to measure cognitive function; and 3) lumbar punctures to obtain CSF samples, which are used to determine the pharmacokinetics of antiretroviral agents in CSF and to determine levels of blood cells, cytokine and immune activation markers, and HIV-1 RNA and DNA. An entry visit must occur before initiating potent antiretroviral therapy in the parent trial [AS PER AMENDMENT 06/06/00: or before changing the antiretroviral regimen due to virologic failure in an ongoing trial]. [AS PER AMENDMENT 11/15/01: Patients are registered before initiating a new potent antiretroviral regimen.] Subsequent visits occur within 21 days prior to each lumbar puncture and at Weeks 24 and 52. If evaluations, procedures, or assays for a given patient's parent trial [AS PER AMENDMENT 11/15/01: for any coenrollment AACTG study] occur at the times specified in this study, they are not duplicated for this study. Other visits may occur when a patient changes antiretroviral treatment or discontinues a parent trial [AS PER AMENDMENT 11/15/01: discontinues a potent antiretroviral therapy].

ELIGIBILITY:
Inclusion Criteria

* Are HIV-positive.
* Have levels of CD4 cells (immune cells that fight infection) less than 200 cells/mm3 and viral loads (level of HIV in the blood) greater than 2,000 copies/ml or viral loads greater than 50,000 copies/ml and any CD4 cell levels.
* Are either: 1) starting a new potent antiretroviral therapy for HIV; 2) enrolling in a potent antiretroviral trial; or 3) currently participating in an ongoing antiretroviral trial or in clinical care and will be changing treatment due to treatment failure. The entry visit for ACTG 736 must occur before starting the treatment or before changing to the new treatment. (This study has been changed to include patients who have changed treatment due to treatment failure and those who are starting a new anti-HIV regimen.)

Exclusion Criteria

* Have an infection or cancer in the brain or certain diseases of the brain or nervous system.
* Have a serious psychiatric illness (such as schizophrenia or severe depression).
* Have completed treatment for a significant infection within 4 weeks of beginning the study (but certain drugs that fight infection are allowed on this study).
* Are taking drugs to prevent or dissolve blood clots.
* Abuse drugs or alcohol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Christina Marra, MD, Study Chair — University of Washington; Kevin Robertson, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (26):
- United States (25):
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Julio Arroyo, West Columbia, South Carolina
  - Comprehensive Care Clinic, Nashville, Tennessee
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico